CLINICAL TRIAL: NCT00382252
Title: Study of Positron Emission Tomography/CT Scan for Response Evaluation After Radiofrequency Ablation in Patients With Lung Metastases
Brief Title: PET Scan and CT Scan in Evaluating Response in Patients Undergoing Radiofrequency Ablation for Lung Metastases
Acronym: TEPARF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000510046; IB-2005-30; INCA-RECF0142; IB-TEP-ARF-MPs-05
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Results first posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Metastatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; lung metastases
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Magnetic Resonance Spectroscopy; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-FDG PET/CT + RFA (Experimental): 18F-FDG PET/CT: I.V. injection of 5 to 15 mCi (185 to 555 MBq) of 18F-FDG. Capture time of 60 to 90 minutes. Acquisition of images: A whole body CT scan with normal breathing will be performed for attenuation correction with 5mm thick slices. A whole body PET acquisition of 6 or 7 steps will be done from the upper third of the thighs to the base of the skull. PETC/CT performed at inclusion, 1 month et 3 months after RFA.
  RFA: Treatment procedure: the location under scanner allows to place the electrode in the center of the tumor. The treatment then lasts 15 to 20 minutes.
  CT scanner: The CT examination will be performed in spiral acquisition without or after injection of contrast medium (70 ml at 2 or 3 ml/sec). On a 16-slice scanner, the examination is performed with 1.25 mm slices every 0.9. Constants generally used 120kV, 350 mA. Ct scanner performed at inclusion, 48H post-RFA, 1 month, 3 months, 6, 9 and 12 months after RFA.
  Interventions: Procedure: computed tomography; Procedure: positron emission tomography; Procedure: radiofrequency ablation

INTERVENTIONS:
Procedure: computed tomography
Procedure: positron emission tomography
Procedure: radiofrequency ablation

SUMMARY:
RATIONALE: Radiofrequency ablation uses a high-frequency, electric current to kill tumor cells. Diagnostic procedures, such as PET scan and CT scan, may help doctors measure the patient's response to treatment.

PURPOSE: This clinical trial is studying PET scan and CT scan to see how well they work in evaluating response to treatment in patients undergoing radiofrequency ablation for lung metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the accuracy of positron emission tomography (PET) and CT scan in measuring response at 3 months after radiofrequency ablation (RFA) in patients with lung metastases.

Secondary

* Determine the agreement between observers analyzing PET/CT scan results.
* Determine the outcome of these patients.
* Determine the false-positive rate and false-negative rate of PET/CT scan at 1 and 3 months in these patients.
* Determine the optimal time for obtaining a negative PET scan.
* Determine the sensitivity, specificity, positive predictive value, and negative predictive value of PET/CT scan at 1 and 3 months.
* Determine the morbidity associated with RFA.
* Determine the disease-free survival after RFA and the factors predicting recurrent disease in these patients.

OUTLINE: This is a multicenter study.

Patients undergo positron emission tomography (PET) and CT scan at baseline. Patients then undergo radiofrequency ablation (RFA) for lung metastases. PET/CT scan is repeated at 1 week, 1 month, and 3 months after RFA.

After completion of RFA, patients are followed by clinical examination and conventional scanning at 6, 9, and 12 months.

PROJECTED ACCRUAL: A total of 80 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed cancer
* Radiologically suspected pulmonary metastases

  * May be confirmed histologically or by specific markers
  * Less than 6 lesions
  * Lesions < 40 mm
  * Prior positron emission tomography shows 1 hyperfixation (standard uptake variable > 3) at the level of lesions to be treated
  * Lesions must not be attached to or next to major mediastinal structures
* Radiofrequency ablation planned as treatment

PATIENT CHARACTERISTICS:

* Life expectancy > 6 months
* No uncontrolled medical condition, including any of the following:

  * Psychiatric condition
  * Infection
  * Coronary insufficiency
  * New York Heart Association class III-IV heart disease
* No other serious condition
* No contraindication to general anesthesia
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

* At least 30 days since prior participation in an investigational study
* At least 30 days since prior chemotherapy
* No other concurrent investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2005-05-02 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francoise Bonichon, MD, Study Chair — Institut Bergonié
Locations (3):
- France (3):
  - Centre Hospitalier de la Cote Basque, Bayonne
  - Institut Bergonie, Bordeaux
  - Hopital Haut Leveque, Pessac

REFERENCES:
- [Derived] Bonichon F, Palussiere J, Godbert Y, Pulido M, Descat E, Devillers A, Meunier C, Leboulleux S, de Baere T, Galy-Lacour C, Lagoarde-Segot L, Cazeau AL. Diagnostic accuracy of 18F-FDG PET/CT for assessing response to radiofrequency ablation treatment in lung metastases: a multicentre prospective study. Eur J Nucl Med Mol Imaging. 2013 Dec;40(12):1817-27. doi: 10.1007/s00259-013-2521-9. Epub 2013 Sep 17. PMID 24042540

RESULTS

PARTICIPANT FLOW:
Groups:
- 18F-FDG PET/CT + RFA: 18F-FDG PET/CT: I.V. injection of 5 to 15 mCi (185 to 555 MBq) of 18F-FDG. Capture time of 60 to 90 minutes. Acquisition of images: A whole body CT scan with normal breathing will be performed for attenuation correction with 5mm thick slices. A whole body PET acquisition of 6 or 7 steps will be done from the upper third of the thighs to the base of the skull. PETC/CT performed at inclusion, 1 month et 3 months after RFA.
  RFA: Treatment procedure: the location under scanner allows to place the electrode in the center of the tumor. The treatment then lasts 15 to 20 minutes.
  CT scanner: The CT examination will be performed in spiral acquisition without or after injection of contrast medium (70 ml at 2 or 3 ml/sec). On a 16-slice scanner, the examination is performed with 1.25 mm slices every 0.9. Constants generally used 120kV, 350 mA. Ct scanner performed at inclusion, 48H post-RFA, 1 month, 3 months, 6, 9 and 12 months after RFA.
  computed tomography
  positron emission tomography
  radiofrequency ablation
Period: Overall Study
Arm/Group | 18F-FDG PET/CT + RFA
Started | 89
Completed | 76
Not Completed | 13
Not completed — Death | 4
Not completed — Protocol Violation | 8
Not completed — Not treated by RFA | 1

BASELINE CHARACTERISTICS:
Arm/Group | 18F-FDG PET/CT + RFA
Number analyzed (Participants) | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 2 patients for whom sex was not available
  Participants
    number analyzed (Participants) | 87
    Female | 41
    Male | 46
Region of Enrollment [Number; unit: participants]
  France | 89

OUTCOME MEASURES:

1. Primary Outcome: Percentage of True Positive Plus True Negative Patients
Description: Accuracy of PET/CT scan to determine response of patients at 3 months will be assessed and compared with standard biopsy 3 months after RFA ,if performed or follow-up at 12 months.
  Number of patients with true positive results plus number of patients with true negative results divided by the number of evaluable patients (accuracy).
Time Frame: 3 months after RFA
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 18F-FDG PET/CT + RFA
Number analyzed (Participants) | 76
percentage of participants | 40.79 [29.65 to 52.67]

2. Secondary Outcome: Percentage of True Positive Patients
Description: Sensitivity of PET/CT scan to determine response of patients at 3 months will be assessed and compared with standard biopsy 3 months after RFA ,if performed or follow-up at 12 months.
  Number of patients with true positive results divided by the number of patients with true positive plus false negative results (sensitivity)
Time Frame: 3 months after RFA
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 18F-FDG PET/CT + RFA
Number analyzed (Participants) | 76
percentage of participants | 100 [69.15 to 100]

3. Secondary Outcome: Percentage of True Negative Patients
Description: Specificity of PET/CT scan to determine response of patients at 3 months will be assessed and compared with standard biopsy 3 months after RFA ,if performed or follow-up at 12 months.
  Number of patients with true negative results divided by the number of patients with true negative plus false positive results (specificity)
Time Frame: 3 months after RFA
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 18F-FDG PET/CT + RFA
Number analyzed (Participants) | 76
percentage of participants | 31.82 [20.89 to 44.44]

ADVERSE EVENTS:
Description: Only serious adverse events were monitored. Adverse events (non-serious) were not assessed/monitored during the study.
Arm/Group | 18F-FDG PET/CT + RFA
Serious Adverse Events (participants affected / at risk) | 2/89
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 18F-FDG PET/CT + RFA (N=89)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes